CLINICAL TRIAL: NCT00780481
Title: Characterization of Brachial Arterial t-PA Release, Vasodilator Function, and Vascular Compliance and Correlation With Fibrinolytic Balance, Oxidative Stress, and Inflammation Measures (SCCOR Project 1 Aim 3B)
Brief Title: Characterization of Brachial Arterial t-PA Release, Endothelial Function, Obesity and Inflammation
Acronym: P1A3B
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment due to strict inclusion/exclusion criteria. Bradykinin shortage
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 061160
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Obesity; Endothelial Function; Fibrinolytic Balance; Baseline
MeSH Terms: conditions — Obesity | interventions — Bradykinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bradykinin (Experimental): Patients will have flow mediated vasodilation and radial artery tonometry performed. They will then receive 0, 10, 20, 40 ng/100cc/min of intrabrachial bradykinin. Strain gauge plethysmography and blood sampling at each dose will be done to evaluate t-PA release. Blood will also be drawn for other biomarkers.
  Interventions: Drug: Bradykinin

INTERVENTIONS:
Drug: Bradykinin — Intrabrachial - 0, 10, 20, 40 ng/100cc/min over 5 minutes at each dose.

SUMMARY:
T-PA release is impaired in obese subjects. In order to have a better mechanistic understanding of t-PA release, we will compare t-PA release to Flow Mediated Vasodilation, Radial Artery Tonometry, and other markers of endothelial function and oxidative stress.

ELIGIBILITY:
Inclusion criteria:

1. Adults 18 years and greater
2. Healthy

Exclusion criteria:

1. PVC < 30
2. Hypertensive subjects on ACE inhibitors
3. Pregnant or nursing mothers
4. Diabetic with HbA1C > 7.5 or stigmata of end organ damage (neuropathy, retinopathy, nephropathy, cardiomyopathy)
5. Cholesterol > 30 mg/dL above NCEP accepted level based on cardiac risk.
6. Triglycerides > 200
7. Previously diagnosed obstructive coronary artery disease, myocardial infarction or left ventricular dysfunction (with or without a history of congestive heart failure)
8. Renal insufficiency (Creatinine ≥ 1.5 mg/dl)
9. History of cerebrovascular disease
10. Any chronic inflammatory disease (rheumatologic, inflammatory bowel disease, etc)
11. Uncontrolled Stage 2 Hypertension (160/100 mmHg), or end organ damage due to hypertension (left ventricular hypertrophy, atrial fibrillation, hematuria, renal insufficiency, prior cerebrovascular disease).
12. Angiotensin converting enzyme inhibitor use
13. Coagulopathy (INR ≥ 1.5, PTT ≥ 1.5 x control)
14. Other chronic medical illnesses at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James AS Muldowney, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data for this study was lost. The total number of participants enrolled/completed was pulled from IRB records. Participant age was between 18-65 per protocol. All participants were enrolled in the United States. No other data is available
Period: Overall Study
Arm/Group | Bradykinin
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data was lost, we do not have sex/gender
Arm/Group | Bradykinin
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: NA: Data was lost
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Peak t-PA Release
Description: tPA Release
Time Frame: Single Study day
Population: Data was lost
Arm/Group | Bradykinin
Number analyzed (Participants) | 0

2. Secondary Outcome: Peak FMD
Time Frame: Single Study Day
Population: Data Lost
Arm/Group | Bradykinin
Number analyzed (Participants) | 0

3. Secondary Outcome: Radial Artery Elasticity
Time Frame: Single Study Visit
Population: Data was lost
Arm/Group | Bradykinin
Number analyzed (Participants) | 0

4. Secondary Outcome: Lipid Levels, PAI-1 Levels, CRP Levels, F2 Isoprostanes and Other Biomarkers of Inflammation and Obesity.
Time Frame: Single Study Day
Population: Data was lost
Arm/Group | Bradykinin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: All data for this study was lost. Unable to provide any information on adverse events.
Arm/Group | Bradykinin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No